CLINICAL TRIAL: NCT05909839
Title: The STEREO-DBS Study: 7-Tesla MRI Brain Network Analysis for Deep Brain Stimulation in Essential Tremor
Brief Title: The STEREO-DBS ET Study: 7-Tesla MRI Brain Network Analysis for Deep Brain Stimulation in Essential Tremor
Acronym: STEREO-ET
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Maarten Bot, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_056 # 21.062
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
Keywords: Brain diseases; Deep brain stimulation; Humans
MeSH Terms: conditions — Essential Tremor; Brain Diseases | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 7T MRI network analysis for deep brain stimulation in essential tremor — We hypothesize that the implementation of 7T MRI network analysis can enhance the effectiveness of DBS by improving motor symptoms and quality of life in ET patients.

SUMMARY:
Rationale: Deep brain stimulation (DBS) of the thalamus is an effective surgical treatment for the patients with advanced essential tremor, despite optimal pharmacological treatment. However, individual improvement after DBS remains variable and 20% of patients experience side effects. To date, DBS-electrode placement and settings in the highly connected thalamus are based on 1,5-Tesla or 3-Tesla MR-images. These low resolution and solely structural modalities are unable to visualize the multiple brain networks to this small nucleus and prevent electrode activation directed at its cortical projections. By using structural 7-Tesla MRI (7T MRI) connectivity to visualize (malfunctioning) brain networks, DBS-electrode placement and activation can be individualized.

Objective: Primary objective of the study is to determine whether visualisation of cortical projections originating in the thalamus and the position of the DBS electrode relative to these projections using 7T MRI improves tremor as measured by the clinically validated Essential Tremor Rating Assessment Scale after six months of DBS.

Secondary outcomes are: disease related daily functioning, adverse effects, operation time, quality of life, patient satisfaction with treatment outcome and patient evaluation of treatment burden.

Study design: The study will be a single center prospective observational study.

Study population: Enrollment will be ongoing from June 2023. Intervention (if applicable): No intervention will be applied. Application of 7T MRI for DBS is standard care and outcome scores used will be readily accessible from the already existing advanced electronic DBS database.

Main study parameters/endpoints: The primary outcome measure is the change in motor symptoms as measured by the disease-specific Essential Tremor Rating Assessment Scale (TETRAS). This is measured after 6 months of DBS as part of standard care. The secondary outcome measures are the Amsterdam Linear Disability Score for functional health status, Quality of Life in Essential Tremor Questionnaire, patient satisfaction with the treatment, patient evaluation of treatment burden, operating time, hospitalization time, change of tremor medication, side effects and complications.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The proposed observational research project involves treatment options that are standard care in daily practice. The therapies will not be combined with other research products. Participation in this study constitutes negligible risk according to NFU criteria for human research.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Deep brain stimulation (DBS) is an effective treatment in essential tremor (ET), a slowly progressive neurological disorder. The effect of DBS relies on the modulation of malfunctioning brain networks by delivering electrical pulses within the thalamus. However, individual improvement after DBS remains variable and 20% of patients experience side effects. By using structural 7-Tesla magnetic resonance imaging (7T MRI) connectivity to visualize malfunctioning networks, DBS-electrode placement and activation can be individualized.

Current DBS-electrode placement and settings in the highly connected thalamus are based on 1.5-Tesla or 3-Tesla MR-images. These low resolution modalities are unable to visualize the multiple brain networks to this small nucleus and prevent electrode activation directed at its cortical projections. Integrated structural (7T MRI) network maps will enable brain network-based and patient-specific DBS, improving motor symptoms and quality of life.

Since the 1980s, DBS for ET was targeting the thalamus, a deep-seated grey matter brain nucleus. Current emphasis in the field of DBS is on neural networks rather than separate nuclei in the brain. Several studies showed ET to arise from pathological network activity in cerebellar-thalamic-cortical projections; dentato-rubro-thalamic-tract. In recent years several DBS groups reported about using MRI to visualize thalamic connectivity and the dentato-rubro-thalamic tract, in DBS for ET.

The thalamus is part of multiple large brain networks. DBS is effective in improving tremor and quality of life for ET patients only by modulating its motor network. For improving DBS placement and activation, it is essential to understand the networks and the modulatory effect of stimulation. Thus far, visualization of these networks was limited due to low resolution and the lack of structural connectivity (visualising -cerebellar-thalamic-cortical projections using diffusion weighted MRI and probabilistic connectivity).

The investigators therefore added 7T T2, FGATIR (fast gray matter inversion recovery sequence) and diffusion-weighted sequences at the Spinoza Centre and showed that probabilistic thalamic network analyses (thalamic segmentation) successfully identifies the area within the thalamus that has the highest density of connections with the motor network in ET patients. In a recent pilot study the investigators showed the implementation of 7T MRI thalamic segmentation is well suited within the existing surgical workflow. By generating a 7-Tesla MRI showing the thalamus (coloured) motor subdivision, this technique clearly visualized this new DBS target.

The thalamus and its connections will be visualized using 7T T2, FGATIR and diffusion weighted imaging. The major projections of the thalamus will be visualised, including projections connecting to primary motor and sendory cortex. The location of the electrode (using computed tomography) will be visualised relative to the segmented subdivisions of the thalamus.

The 7T MRI network map, generated by combining T2 and diffusion weighted MRI, shows the thalamus (coloured) subdivisions and their cortical projections. The result will then show in which thalamic subdivision(s) the DBS-electrode contact is situated and to which cortical area this projects. Clinical test scores of the electrode contact will then be correlated to the network maps. Stimulation parameters based on 7T MRI network maps are used to optimize and predict outcome in terms of beneficial clinical effects (suppression tremor) and side effects (speech, gait). As all network maps are visualised on MRI, this will readily enable both individual and group analyses (co-registrating maps of multiple patients).

In the 350 7T MR-scans the investigators have performed to date, we rarely encountered non-compatible implants or severe claustrophobia. Every patient undergoes screening with a MRI safety questionnaire and MRI metal detector (preventing taking ferromagnetic materials into the MRI). 7T MRI is a non-invasive technique which causes no pain and, importantly, the electromagnetic fields produce no known tissue damage of any kind. The MR system may make loud tapping, knocking, or other noises at times during the procedure. Earplugs are provided to prevent problems that may be associated with noise generated by the scanner. At all times, the patient will be (visually) monitored and will be able to communicate with the 7T MRI technologist using an intercom system. The patient may (request to) stop the acquisition at any time by using the push button (hold by the patient continuously).

In sum, due to implementation of 7T MRI brain network analysis, it is now possibly to directly visualize the motor part of the thalamus. In current observational study this technique will be evaluated in a prospective fashion, introducing patient specific brain network-guided DBS for ET with delivering a unique and hitherto unavailable treatment and dataset: 7T MRI visualizes the anatomical connections of the thalamus for each individual DBS electrode contact. Instead of a one-brain-fits all model, the tailored network analyses enable personalized precision modelling in DBS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Idiopathic essential tremor who underwent DBS

Exclusion Criteria:

* Legally incompetent adults
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced essential tremor who underwent DBS electrode placement using 7T MRI network analysis. If the patient is eligible, the physician coordinating the study will inform the patient, hand over written information about the observational study, and subsequently ask the patient to consider participation. If the patient wants to participate, the informed consent form will be signed. Patients will be given as much time as needed to decide whether to participate in the study. Enrollment will be ongoing from June2023; patients who underwent 7T MRI network analysis based DBS before this date will also be eligible to participate (all DBS patients are registered in the prospective electronic Castor database).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2033-06-09 (Estimated); Study Completion 2033-06-09 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Rating Assessment Scale (TETRAS) | June 2023 - June 2033
  The amount of decrease in motor symptoms indicated by change in the disease-specific Essential Tremor Rating Assessment Scale (TETRAS) after six months of deep brain stimulation. The TETRAS scores are between 0 and 64; higher scores indicating worse (more severe) tremor symptoms.

SECONDARY OUTCOMES:
The Amsterdam Linear Disability Score for functional health status | June 2023 - June 2033
  The Amsterdam Linear Disability Score (ALDS) is a generic itembank which measures disability, as expressed by the ability to perform activities of daily living. These scores are linearly transformed into values between 0 and 100. Lower scores indicate more disability.
Quality of Life in Essential Tremor Questionnaire | June 2023 - June 2033
  The Quality of Life in Essential Tremor Questionnaire (QUEST) is a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL) that generic QOL measures do not effectively capture, including activities of daily living that are affected by essential tremor. The QUEST was made to be relatively brief and easy for patients to use.
Global Impression of Change | June 2023 - June 2033
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI actually comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale.
EQ-5D-5L | June 2023 - June 2033
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting june 2023
Access Criteria: open access

REFERENCES:
- [Background] 1. Song P, Zhang Y, Zha M, et al. The global prevalence of essential tremor, with emphasis on age and sex: A meta-analysis. J Glob Health. Apr 10 2021;11:04028. 2. Schuurman PR, Bosch DA, Merkus MP, Speelman JD. Long-term follow-up of thalamic stimulation versus thalamotomy for tremor suppression. Movement disorders : official journal of the Movement Disorder Society. Jun 15 2008;23(8):1146-1153. 3. Bot M, van Rootselaar F, Contarino MF, et al. Deep Brain Stimulation for Essential Tremor: Aligning Thalamic and Posterior Subthalamic Targets in 1 Surgical Trajectory. Oper Neurosurg (Hagerstown). Aug 1 2018;15(2):144-152. 4. Bot M, van Rootselaari AF, Odekerken V, et al. Evaluating and Optimizing Dentato-Rubro-Thalamic-Tract Deterministic Tractography in Deep Brain Stimulation for Essential Tremor. Oper Neurosurg (Hagerstown). Sep 25 2021. 5. Bot M, Pauwels R, van den Munckhof P, et al. The Fast Gray Matter Acquisition T1 Inversion Recovery Sequence in Deep Brain Stimulation: Introducing the Rubral Wing for Dentato-Rubro-Thalamic Tract Depiction and Tremor Control. Neuromodulation. Jan 15 2022. 6. Holewijn RA, Verbaan D, van den Munckhof PM, et al. General Anesthesia vs Local Anesthesia in Microelectrode Recording-Guided Deep-Brain Stimulation for Parkinson Disease: The GALAXY Randomized Clinical Trial. JAMA Neurol. Sep 7 2021. 7. Graat I, Mocking RJT, Liebrand LC, et al. Tractography-based versus anatomical landmark-based targeting in vALIC deep brain stimulation for refractory obsessive-compulsive disorder. Mol Psychiatry. Dec 2022;27(12):5206-5212. 8. Nowacki A, Barlatey S, Al-Fatly B, et al. Probabilistic Mapping Reveals Optimal Stimulation Site in Essential Tremor. Ann Neurol. May 2022;91(5):602-612. 9. Coenen VA, Sajonz B, Prokop T, et al. The dentato-rubro-thalamic tract as the potential common deep brain stimulation target for tremor of various origin: an observational case series. Acta neurochirurgica. May 2020;162(5):1053-1066. 10. Akram H, Dayal V, Mahlknecht P, et al. Connectivity derived thalamic segmentation in deep brain stimulation for tremor. Neuroimage Clin. 2018;18:130-142. 11. Nowacki A, Schlaier J, Debove I, Pollo C. Validation of diffusion tensor imaging tractography to visualize the dentatorubrothalamic tract for surgical planning. Journal of neurosurgery. Mar 23 2018;130(1):99-108. 12. Coenen VA, Allert N, Paus S, Kronenburger M, Urbach H, Madler B. Modulation of the Cerebello-Thalamo-Cortical Network in Thalamic Deep Brain Stimulation for Tremor: A Diffusion Tensor Imaging Study. Neurosurgery. Dec 2014;75(6):657-669. 13. Kremer NI, Pauwels RWJ, Pozzi NG, et al. Deep Brain Stimulation for Tremor: Update on Long-Term Outcomes, Target Considerations and Future Directions. J Clin Med. Aug 5 2021;10(16).